CLINICAL TRIAL: NCT01897805
Title: A Randomized, Double-blind, Multi-centered, Placebo-controlled Trial to Examine Effects of Heart-protecting Musk Pill on Clinical Outcome in Patients With Chronic Stable Coronary Artery Disease
Brief Title: A Trial to Evaluate Efficacy of Heart-protecting Musk Pill
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Hutchison Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG0930BXW
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heart-protecting Musk Pill (Experimental): Patients will get standard treatment for coronary artery disease plus 2 Heart-protecting Musk Pills each time, three times a day by mouth for 24 months
  Interventions: Drug: Heart-protecting Musk Pill
- Placebo (Placebo Comparator): Patients will get standard treatment for coronary artery disease plus 2 placebo pills each time, three times a day by mouth for 24 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Heart-protecting Musk Pill
  Arms: Heart-protecting Musk Pill
Drug: Placebo
  Arms: Placebo

SUMMARY:
Title:

A randomized, double-blind, multi-centered, placebo-controlled trial to examine effects of of Heart-protecting Musk Pill on clinical outcomes in patients with chronic stable coronary artery disease

Objective:

To examine effects of of Heart-protecting Musk Pill, a traditional Chinese medicine, on clinical outcomes in patients with chronic stable coronary artery disease

The study hypothesis:

The null hypothesis: the combined incidence of cardiovascular death, nonfatal myocardial infarction, nonfatal stroke in the treatment group is the same as that in control group.

The alternative hypothesis: the combined incidence of cardiovascular death, nonfatal myocardial infarction, nonfatal stroke in the treatment group is different from that in control group.

Sample size:

2700 patients will be randomized, 1350 in treatment group and 1350 in placebo group.

Number of sites: 99 sites in China

Study drugs:

Heart-protecting Musk Pill and the matching placebo pills.

Design:

A randomized, double-blind, multi-centered, placebo-controlled trial. Patients will be randomized to treatment group and placebo group after screening and get corresponding treatment as follow.

Treatment group: Standard treatment for coronary artery disease plus 2 Heart-protecting Musk Pills each time, three times a day by mouth for 24 months.

Control group: Standard treatment for coronary artery disease plus 2 placebo pills each time, three times a day by mouth for 24 months.

Patients will be followed up at baseline, 1, 3, 6, 9, 12, 18, 24 months after randomization. During follow-up period, patients could undertake PCI or CABG if angina get out of control or evidence of ischemia aggravated is found.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years at screening.
2. Patients who have ischemia myocardial symptoms and whose clinical symptoms keep stable for at least one month.
3. Have at least one of the following events (providing hospital records or inspection report): 1)history of acute myocardial infarction for at least half of a year; 2) history of PCI or CABG for at least half of a year; 3) coronary CT angiography or coronary angiography shows that at least one of the main branches of coronary artery stenosis is no less than 50%.
4. Provide informed consent form.

Exclusion Criteria:

1. History of acute myocardial infarction, vascular reconstruction, CABG or PCI within half of a year.
2. Prepared to undertake CABG or PCI during this study.
3. Serious cardiovascular diseases: sustained severe angina (CCS Ⅳ), refractory heart failure, cardiogenic shock, severe aortic stenosis or aortic insufficiency.
4. Severe respiratory diseases;
5. Diabetic patients with poor glycemic control (fasting blood glucose > 200 mg/dl or 11.1mmol/L for more than twice within one month before the study entry).
6. Hypertensive patients with poor control of blood pressure, systolic pressure≥180mmHg or diastolic pressure≥110mmHg before entry.
7. Severe liver and kidney diseases,such as active liver disease, cirrhosis and uremia.
8. Any other severe diseases, such as malignant tumor, severe anemia and severe renal artery stenosis.
9. Unable or unwilling to sign informed consent form.
10. Join another trial or has received random allocation of this study within one month before entry.
11. Pregnant or who were attempting to become pregnant.
12. Patients who are regarded as not being suitable participants by the study investigators.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2700 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The combined incidence of cardiovascular death, nonfatal myocardial infarction, nonfatal stroke | 24 months

SECONDARY OUTCOMES:
The combined incidence of all-cause mortality, nonfatal myocardial infarction, nonfatal stroke, hospitalization for unstable angina or heart failure, and peripheral revascularization (PCI or CABG) | 24 months

OTHER OUTCOMES:
The incidence of adverse event | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Doctor, Principal Investigator — Fudan University
Locations (98):
- China (98):
  - AnHui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Medical University Of Anhui, Hefei, Anhui
  - MaAnShan Central Hospital, Maanshan, Anhui
  - Beijing An Zhen Hospital of the Capital University of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital Capital Medical University, Beijing, Beijing Municipality
  - Dongfang Hospital Affiliated to Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Navi General Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Armed police Chongqing Corps Hospital, Chongqing, Chongqing Municipality
  - The Third People's Hospital of Chongqing, Chongqing, Chongqing Municipality
  - FuJian Provincial Hospital, Fuzhou, Fujian
  - People's Hospital of Fujian Province, Fuzhou, Fujian
  - The Affiliated Hospital of PuTian University, Putian, Fujian
  - XiaMen Heart Center, Xiamen, Fujian
  - Affiliated Hospital of Guangzhou Medcal College, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - The First Affiliated Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - The People's Hospital of Jiangmen, Jiangmen, Guangdong
  - ShenZhen People's Hospital, Shenzhen, Guangdong
  - The Affiliated Hospital of Guangdong Medical College, Zhanjiang, Guangdong
  - The First People's Hospital of Liuzhou City, Liuchow, Guangxi
  - The First Affiliated Hospital Of GuangXi University Of Chinese Medicine, Nanning, Guangxi
  - HeBei General Hosital, Shijiazhuang, Hebei
  - The Seond Hospital of HeBei Medical University, Shijiazhuang, Hebei
  - TangShan GongRen Hospital, Tangshan, Hebei
  - DaQing General Hospial Group LongNan Hosptial, Daqing, Heilongjiang
  - KaiFeng Central Hospital, Kaifeng, Henan
  - People's Hospital of Henan Province, Zhengzhou, Henan
  - The First Affiliated Hospital of Henan University of TCM, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Affiliated Hospital of Henan University of TCM, Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Taihe Hospital, Shiyan, Hubei
  - Hubei Provincial Corps Hospital of CPAPF, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The First People's Hospital of Changde, Changde, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central-South University, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - JiangSu Province Hosptial of TCM, Nanjing, Jiangsu
  - JiangSu Province Hosptial, Nanjing, Jiangsu
  - NanJing Drum Tower Hospital The Affiliated Hospital of NanJing University Medical School, Nanjing, Jiangsu
  - NanJing First Hospital, Nanjing, Jiangsu
  - NanJing Hospital of TCM, Nanjing, Jiangsu
  - SuZhou Municipal Hospital, Suzhou, Jiangsu
  - JiangSu TaiZhou People's Hospital, Taizhou, Jiangsu
  - WuXi People's Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of XuZhou Medical College, Xuzhou, Jiangsu
  - Northern JiangSu People's Hospital, Yangzhou, Jiangsu
  - YangZhou No. 1 People's Hospital, Yangzhou, Jiangsu
  - The Affiliated Hospital of JiangXi University of Traditional Chinese Medicine, Nanchang, Jiangxi
  - The First Hospital of NanChang, Nanchang, Jiangxi
  - The Second Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The First Hospital Of China Medical University, Anshan, Liaoning
  - The 210th Hospital of Chinese people's Liberation Army, Dalian, Liaoning
  - The second people's Hospital of Dalian, Dalian, Liaoning
  - Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Affiliated Hospital of Shandong University of TCM, Jinan, Shandong
  - Shangdong Provincial Hospital, Jinan, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Qilu Hospital of Shandong University, Qinan, Shandong
  - Qingdao University Medical College Affiliated Yuhuangding Hospital, Qingdao, Shandong
  - The Affiliated Hospital of Medical College of Qingdao University, Yantai, Shandong
  - Huadong Hospital Affiliated To Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Shuguang Hospital, Shanghai, Shanghai Municipality
  - Tongji Hospital Affiliated to Tongji University, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Medical University First Hospital, Taiyuan, Shanxi
  - Shanxi Medical University Second Hospital, Taiyuan, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Affiliated Hospital of Luzhou Medical College, Luzhou, Sichuan
  - Affiliated Hospital of Chuanbei Medical College, Nanchong, Sichuan
  - The First Teaching Hospital of TianJin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - TianHe Hospital, Tianjin, Tianjin Municipality
  - TianJin Chest Hospital, Tianjin, Tianjin Municipality
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Yunnan Provincial Hospital of Traditional Chinese Medicine, Kunming, Yunnan
  - Hangzhou Traditional Chinese Medical Hospital, Hangzhou, Zhejiang
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - The First Affiliated Hospital ZheJiang University, Hangzhou, Zhejiang
  - Tongde Hospital of ZheJiang Province, Hangzhou, Zhejiang
  - ZheJiang Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial Hospital of TCM, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Ningbo Medical Treatment Center of LiHuiLi Hospital, Ningbo, Zhejiang
  - The Second Hospital Affiliated to Wenzhou Medical College, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Shi H, Zhou J, Ma C, Ji F, Wu Y, Zhao Y, Qian J, Wang X. Shexiang Baoxin Pill (MUSKARDIA) reduces major adverse cardiovascular events in women with stable coronary artery disease: A subgroup analysis of a phase IV randomized clinical trial. Front Cardiovasc Med. 2022 Oct 21;9:1002400. doi: 10.3389/fcvm.2022.1002400. eCollection 2022. PMID 36386372